CLINICAL TRIAL: NCT01472094
Title: Clinical and Biological Predictors of Chemotherapy Toxicity in Older Adults
Brief Title: The Hurria Older PatiEnts (HOPE) With Breast Cancer Study
Status: Active, not recruiting | Type: Observational
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: 11127; 1R01AG037037-01 (NIH)
Record Dates: First submitted 2011-10-31; First posted 2011-11-16 (Estimated); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients: All patients 65 years old with Stage I to III breast cancer who are beginning adjuvant or neo-adjuvant chemotherapy.

SUMMARY:
The goal of this study is to develop a "bedside to bench" model of clinical and biological predictors for toxicity to adjuvant and neoadjuvant chemotherapy in older adults with breast cancer. The investigators will develop a predictive model using clinical and biological predictors of toxicity to adjuvant and neoadjuvant chemotherapy in older adults with breast cancer. The investigators will also determine the association between clinical and biological factors and reduced relative dose intensity of the prescribed chemotherapy regimen. In addition, the investigators will explore specific chemotherapy toxicities associated with reduced relative dose intensity of a prescribed regimen.

DETAILED DESCRIPTION:
Although cancer is a disease associated with aging, there is no standard tool in oncology practice that incorporates clinical and biological factors to identify older adults with cancer who may be more vulnerable to the toxicity of chemotherapy. It is generally recognized that chronological age tells relatively little about an older adult's physiological age. Oncologists allude to this when they describe an older adult as: "a 'young' 80-year-old" or "an 'old' 80-year-old," implying factors other than age contribute to the health status of an older adult. Geriatricians address this by routinely performing a "geriatric assessment," which measures independent clinical predictors of morbidity and mortality in older adults. In addition, several potential biomarkers of aging have been described that are associated with functional decline and mortality among older adults. This study will identify whether novel biomarkers of aging can predict risk of chemotherapy toxicity. The current proposal will fill this knowledge gap by melding the principles of geriatrics with those of oncology to create a tool to assess the clinical and biological risk factors for chemotherapy toxicity in older adults.

Furthermore, this study will determine the association between chemotherapy toxicity and dose reductions and/or delays that decrease chemotherapy dose intensity. Maintenance of chemotherapy dose intensity is necessary to maintain chemotherapy efficacy. Older adults are at risk for chemotherapy toxicity and if this toxicity results in decreased dose intensity, the benefits of chemotherapy will be compromised. This study will identify the association between clinical and biological predictors of grade 2-5 toxicity and relative dose intensity. Furthermore, this study will identify the specific dose-limiting toxicities. These data will provide evidence-based criteria to identify those patients whose projected risk of toxicity would limit dose intensity and compromise the efficacy of standard treatment. These data could serve as the basis for "vulnerable elderly trials" which would study an alternate therapy regimen in patients who are predicted to have a significant risk of toxicity (and compromised efficacy) with the standard regimen.

This proposal unites the fields of geriatrics and oncology, incorporating geriatric correlates of vulnerability and studying their impact in an aging oncology population. These data will be used to develop a predictive equation for the risk of chemotherapy toxicity that can be utilized in daily oncology practice. These data will facilitate decision-making regarding the risks and benefits of adjuvant chemotherapy in older adults with breast cancer and ultimately serve as a foundation on which to identify older adults at risk for chemotherapy toxicity in order to guide interventions to decrease this risk.

ELIGIBILITY:
Patients with Breast Cancer:

Inclusion Criteria:

* Patients with stages I-III breast cancer receiving adjuvant or neoadjuvant chemotherapy
* Able to understand English
* Able to provide informed consent
* Patients age ≥65 and of any performance status are eligible

Exclusion Criteria:

* Patients with metastatic disease

Breast Cancer Controls:

Inclusion Criteria:

* Patients with stages I-III breast cancer
* Patient will not receive adjuvant or neoadjuvant chemotherapy
* Patients age ≥65 and of any performance status are eligible
* Able to understand English
* Able to provide informed consent

Exclusion Criteria:

* Patients with metastatic disease
* Receipt of chemotherapy

Healthy Controls:

Inclusion Criteria:

* Patients age ≥65 and of any performance status are eligible
* No history of cancer (excluding non-melanoma skin cancer)
* Able to understand English
* Able to provide informed consent

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Outpatient clinic practices (City of Hope, Memorial Sloan-Kettering Cancer Center, Yale University School of Medicine, University of Rochester, University of North Carolina, Wake Forest University, and Case Western Reserve University)
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2011-09-09 (Actual); Primary Completion 2018-12-02 (Actual); Study Completion 2026-09-18 (Estimated)

PRIMARY OUTCOMES:
Develop a predictive model of clinical and biological predictors for grade 2-5 toxicity to adjuvant and neoadjuvant chemotherapy. | 6 months after completion of chemotherapy
Understand the association between clinical and biological factors and reduced relative dose intensity (RDI) of the prescribed chemotherapy regimen. | 6 months after completion of chemotherapy
Identify the specific chemotherapy toxicities associated with reduced relative dose intensity of the prescribed chemotherapy regimen. | 6 months after completion of chemotherapy
Understand the association between the receipt of adjuvant chemotherapy and change in functional status from pre-chemotherapy to end of chemotherapy. | 6 months after completion of chemotherapy

SECONDARY OUTCOMES:
Assess potential biomarkers for physiologic age, including interleukin-6, C-reactive protein, D-dimer, and p16 expression. | 6 months after completion of chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Mina Sedrak, MD, Principal Investigator — City of Hope Medical Center
Locations (17):
- United States (17):
  - City of Hope Medical Center, Duarte, California
  - Yale University, New Haven, Connecticut
  - University of Chicago, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Washington University St. Louis, St Louis, Missouri
  - Roswell Park Cancer Institute, Buffalo, New York
  - Hofstra-North-LIJ Cancer Institute, New Hyde Park, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Wake Forest University, Winston-Salem, North Carolina
  - Case Western Reserve University, Cleveland, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - University of Virginia Health System, Charlottesville, Virginia

REFERENCES:
- [Background] Hurria A, Togawa K, Mohile SG, Owusu C, Klepin HD, Gross CP, Lichtman SM, Gajra A, Bhatia S, Katheria V, Klapper S, Hansen K, Ramani R, Lachs M, Wong FL, Tew WP. Predicting chemotherapy toxicity in older adults with cancer: a prospective multicenter study. J Clin Oncol. 2011 Sep 1;29(25):3457-65. doi: 10.1200/JCO.2011.34.7625. Epub 2011 Aug 1. PMID 21810685
- [Derived] Ji J, Bae M, Sun CL, Wildes TM, Freedman RA, Magnuson A, O'Connor T, Moy B, Klepin HD, Chapman AE, Tew WP, Dotan E, Fenton MA, Kim H, Katheria V, Gross CP, Cohen HJ, Muss HB, Sedrak MS. Falls prechemotherapy and toxicity-related hospitalization during adjuvant chemotherapy for breast cancer in older women: Results from the prospective multicenter HOPE trial. Cancer. 2024 Mar 15;130(6):936-946. doi: 10.1002/cncr.35105. Epub 2023 Nov 14. PMID 37962093
- [Derived] Sedrak MS, Sun CL, Ji J, Cohen HJ, Gross CP, Tew WP, Klepin HD, Wildes TM, Dotan E, Freedman RA, O'Connor T, Chow S, Fenton MA, Moy B, Chapman AE, Dale W, Katheria V, Kuderer NM, Lyman GH, Magnuson A, Muss HB. Low-Intensity Adjuvant Chemotherapy for Breast Cancer in Older Women: Results From the Prospective Multicenter HOPE Trial. J Clin Oncol. 2023 Jan 10;41(2):316-326. doi: 10.1200/JCO.22.01440. Epub 2022 Dec 1. PMID 36455189
- [Derived] Magnuson A, Sedrak MS, Gross CP, Tew WP, Klepin HD, Wildes TM, Muss HB, Dotan E, Freedman RA, O'Connor T, Dale W, Cohen HJ, Katheria V, Arsenyan A, Levi A, Kim H, Mohile S, Hurria A, Sun CL. Development and Validation of a Risk Tool for Predicting Severe Toxicity in Older Adults Receiving Chemotherapy for Early-Stage Breast Cancer. J Clin Oncol. 2021 Feb 20;39(6):608-618. doi: 10.1200/JCO.20.02063. Epub 2021 Jan 14. PMID 33444080
- See also: Related Info — http://www.mycarg.org